CLINICAL TRIAL: NCT04668443
Title: Acceptability and Feasibility of a Graphical Informed Consent in the Informed Consent Process of D²EFT Study
Brief Title: D²EFT Graphical Informed Consent
Acronym: D²EFT-GIC
Status: Completed | Type: Observational
Sponsor: Kirby Institute (Other Government)
Collaborators: Institute of Human Virology, Nigeria (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-02-DEFT-GIC
Record Dates: First submitted 2020-12-03; First posted 2020-12-16 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: HIV-1-infection
Keywords: Informed consent process

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective participants in D²EFT study: HIV-positive persons who are eligible for the D²EFT study will be proposed to receive the research-related information with the set of pictures (GIC)
  Interventions: Other: Graphical Informed Consent (GIC)
- Researchers obtaining informed consent for D²EFT study: Healthcare givers involved in the participant informed consent process of D²EFT
  Interventions: Other: Graphical Informed Consent (GIC)

INTERVENTIONS:
Other: Graphical Informed Consent (GIC) — The GIC (set of illustrations that complement the written information and consent form) will be proposed to prospective participants by researchers, systematically during the pre-test (stage 1). If the stage 1 shows no negative impact of the GIC on the consent process, the stage 2 will be implemented and the GIC will be proposed by researchers when they feel it could be beneficial for the participant.

SUMMARY:
D²EFT-GIC is a substudy of D²EFT study (NCT03017872), a randomised clinical trial of second-line antiretroviral therapies. The goal of D²EFT-GIC is to evaluate a novel tool, the "Graphical Informed Consent" (GIC), within D²EFT.

The GIC is designed to supplement the informed consent process with a set of culturally- and gender-adapted illustrations, with an explanatory script for researchers, that complements the mandatory written participant information sheet and consent form.

The investigators propose to assess the acceptability and feasibility of this tool from the participants and researchers perspectives. The GIC will be first pre-tested in one or more site(s) - where the informed consent process is challenging because of literacy, language or culture barriers - in 10 prospective participants for D²EFT. If this stage shows there is no negative impact of the GIC on the consent process, the second stage will study the feasibility of implementing the GIC in the usual practice.

DETAILED DESCRIPTION:
Informed consent requires provision of complex medical information in an easily understandable format. During the consent process, researchers may encounter potential research participants who are not thoroughly used to care services and thus may struggle to understand what clinical research is, the purpose of the specific research in relation to their health, research methods, its risks and benefits, and their options and rights. Clinical trials in people living with HIV can present additional challenges due to stigma surrounding the infection, as the need for a third-party witness to ensure adequate comprehension of the presented information may be concerning to the participant. These barriers to an optimal informed consent are particularly significant in low and lower-middle income countries (LMICs).

To try to overcome these barriers and to make written information sheet and consent forms (PICFs) more accessible and understandable for key-populations, and more user-friendly for on-site researchers, tools including interactive videos have been developed for various diseases and different settings. Many of these tools are study-specific or developed in high-income countries with limited reproducibility; few have been studied in the consent process for HIV treatment trials or across multiple LMIC settings. Data evaluating these tools and their impact on participants' understanding or researchers' satisfaction are limited.

With the D²EFT community advisory board (CAB) and protocol steering committee (PSC), the investigators developed the "Graphical Informed Consent" (GIC). This tool is designed to supplement the informed consent process with a set of culturally- and gender-adapted illustrations with an explanatory script for researchers, that complement the mandatory written PICF.

The investigators propose to evaluate this novel tool within D²EFT study, a randomised clinical trial of HIV second-line therapy in LMICs, by undertaking a pilot study. The study aims to assess acceptability and feasibility of the GIC by measuring implementation outcomes: participants' acceptability and acceptance, and researchers' utilisation and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Fulfil the eligibility criteria for D²EFT and willing to undertake D²EFT informed consent process;
* Being able to give a verbal consent for the D²EFT-GIC.

Exclusion Criteria:

* Unwilling to comply with the substudy requirements.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective participants for D²EFT study and researchers obtening the informed consent process.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Proportion of prospective D²EFT participants to whom researchers offered the supplemental GIC during the informed consent process (Stage 2) | Up to 1 year
  Utilisation (uptake) of the GIC by researchers: number of times researchers offered the supplemental GIC during the informed consent process of D²EFT divided by the total number of prospective participants who underwent informed consent for D²EFT during the substudy period when the GIC is freely available

SECONDARY OUTCOMES:
Proportion of participants who find the illustrations helpful (Stage 1) | Up to 3 months
  A five-point Likert scale will be used in a questionnaire administered to the participants after they underwent the D²EFT informed consent process with the GIC, during Stage 1. "Overall, supplementing the written information explained by the doctor with illustrations is": multiple answers will range from "Extremely troublesome" (worst outcome) to "Very interesting (helpful)" (best outcome).
Proportion of researchers who think there are issues in using the GIC (Stage 1) | Up to 3 months
  A questionnaire with a three-point Likert scale will be used: "Yes" (worst outcome) to "No" (best outcome).
Proportion of participants who accept to undergo the D²EFT informed consent process with GIC (Stage 2) | Up to 1 year
  Participants' acceptance (uptake) during stage 2. The number of participants who accept/decline the use of illustrations when the researcher offered the GIC with the written informed consent will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Mark Polizzotto, MD, PhD, Principal Investigator — The Kirby Institute, UNSW
Locations (1):
- Institute of Human Virology Nigeria (IHVN), Abuja, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided